CLINICAL TRIAL: NCT01134341
Title: A Phase 1, Open-label, Dose-finding Study of Pralatrexate Plus Systemic Bexarotene in Patients With Relapsed or Refractory Cutaneous T Cell Lymphoma
Brief Title: Pralatrexate and Bexarotene in Patients With Relapsed or Refractory Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-018
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cutaneous T-cell Lymphoma; Mycosis Fungoides; Sezary Syndrome; Primary Cutaneous Anaplastic Large Cell Lymphoma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Recurrence | interventions — 10-propargyl-10-deazaaminopterin; Bexarotene; Vitamin B 12; Folic Acid

ARMS (1):
- Bexarotene (Targretin) & Pralatrexate (Folotyn) (Experimental): Bexarotene (Targretin): administered po qd. The initial daily dose of bexarotene will depend on the cohort to which each patient is assigned. Bexarotene will be self-administered except in patients who underwent plasma PK sampling on cycle 1, dose 1 and cycle 1, dose 3, at which time bexarotene was to be administered at the investigational site 1 hour (± 5 minutes) prior to pralatrexate administration.
  Pralatrexate (Folotyn): administered weekly via IV push over a minimum of 30 seconds up to a maximum of 5 minutes. One cycle is 4 weeks in duration consisting of weekly dosing of pralatrexate for 3 weeks followed by 1 week of rest. The initial dose of pralatrexate will depend on the cohort to which each patient is assigned.
  Interventions: Drug: Pralatrexate Injection; Drug: Bexarotene Capsules; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate Injection — Intravenous (IV) push over 30 seconds to 5 minutes via a patent free-flowing IV line containing normal saline (0.9% sodium chloride).
  10 or 15 mg/m2, depending on cohort assignment.
  Dose reductions allowed for protocol-specified criteria.
  Administered weekly for 3 weeks of 4-week cycle (weekly for 3 weeks with one week of rest) until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; PDX; Pralatrexate; (RS)-10-propargyl-10-deazaaminopterin
Drug: Bexarotene Capsules — 150 or 300 mg orally, depending on cohort assignment. Provided as 75 mg capsules and taken with a meal.
  Dose reductions allowed for protocol-specified criteria and implemented per the Targretin® package insert.
  Administered daily until criteria for study treatment discontinuation per the protocol are met.
  Other Names: Bexarotene; Targretin®
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered within 10 weeks prior to start of study treatment, every 8-10 weeks throughout the study and for 30 days after last study treatment (dose of pralatrexate or bexarotene).
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1-1.25 mg orally
  Administered daily for at least 7 days prior to start of study treatment, throughout the study and for 30 days after last study treatment (dose of pralatrexate or bexarotene).
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
This study is designed to determine the recommended dose, safety, pharmacokinetics, and early efficacy of the combination of pralatrexate plus oral bexarotene in patients with relapsed or refractory CTCL.

DETAILED DESCRIPTION:
This is a multi-center, dose-finding, Phase 1 study of pralatrexate plus bexarotene in patients who have relapsed or refractory CTCL.

Primary Objective(s):

• Determine the maximum tolerated dose (MTD) and recommended dose of pralatrexate plus bexarotene with concurrent vitamin B12 and folic acid supplementation when administered to patients who have failed prior systemic treatment.

Secondary Objective(s):

* Determine the safety profile of pralatrexate plus bexarotene when administered to patients with relapsed/refractory cutaneous T-cell lymphoma (CTCL).
* Collect preliminary efficacy data.
* Determine the pharmacokinetic (PK) profile of pralatrexate plus bexarotene in patients who underwent plasma PK sampling

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous T-cell lymphoma patients with subtypes of mycosis fungoides (MF) Stage IB or higher, Sézary syndrome, or primary cutaneous anaplastic large cell lymphoma who have failed a previous systemic treatment.
* Patients must have received at least 1 previous systemic therapy, and either progressed or not tolerated their last prior treatment regimen.
* Eastern Cooperative Oncology Group Performance Status less than or equal to 2.
* Adequate blood, liver, and kidney function as defined by laboratory tests.
* Women of childbearing potential must practice medically acceptable contraception from study treatment start until at least 30 days after the last dose of study treatment. Negative serum pregnancy test within 14 days before the first day of study treatment (not required for patients who are postmenopausal for at least 1 year or surgically sterilized). Study treatment should not be given to women who are breastfeeding.
* Males who are sexually active must agree to practice medically acceptable barrier contraception while receiving study treatment and for 30 days after the last dose of study treatment.
* Give written informed consent & privacy authorization.

Exclusion Criteria:

* If there is a history of prior malignancies other than non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, or localized thyroid cancer, patient must be disease free for at least 5 years. Patients with other prior malignancies less than 5 years before study entry may be enrolled if they received treatment resulting in complete resolution of the cancer and have no current clinical, radiologic, or laboratory evidence of active or recurrent disease.
* Human immunodeficiency virus (HIV)-positive diagnosis with a CD4 count of less than 100 mm3 or detectable viral load within the past 3 months, and receiving combination anti-retroviral therapy.
* Diagnosis of Hepatitis B virus, or Hepatitis C virus with detectable viral load or immunological evidence of chronic active disease or receiving/requiring antiviral therapy.
* Active central nervous system disease requiring treatment.
* Active uncontrolled infection, underlying medical condition, or other serious illness impairing the patient's ability to receive protocol treatment.
* Discontinuation of prior oral bexarotene due to an allergic reaction or treatment-related toxicity.
* Major surgery within 2 weeks of planned start of treatment.
* Conventional or investigational chemotherapy or radiation therapy encompassing greater than 10% of bone marrow within 4 weeks prior to study treatment.
* ECP, phototherapy with PUVA, or ultraviolet (UV) therapy within 2 weeks prior to study treatment.
* Systemic corticosteroids within 3 weeks of study treatment, unless patient has been taking a continuous dose of no more than 10 mg per day of prednisone or equivalent for at least 4 weeks.
* Initiation of or change in dosage of topical corticosteroids within 3 weeks of study treatment (topical steroid use within 3 weeks is allowed provided the strength and use has been stable for at least 4 weeks).
* Investigational drugs, biologics, or devices use within 2 weeks prior to study treatment or planned use during the study.
* Monoclonal antibody within 3 months without evidence of PD.
* Use of oral retinoids, except bexarotene, within 4 weeks of study treatment or high-dose vitamin A (once daily multi-vitamin allowed).
* Previous exposure to pralatrexate.
* Uncontrolled hypercholesterolemia or hypertriglyceridemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) Rate | Assessed weekly through cycle 1 (weeks 1-4)
  DLT rate is the number of patients experiencing a DLT divided by number of evaluable patients and it will be summarized by dose level.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Assessed after every 2 cycles (8 weeks) for the first 12 months, then every 4 cycles (16 weeks) until progression of disease.
  best overall response is the best response recorded from the start of treatment until PD.
  The objective response rate is the proportion of patients with a best overall response of either CR or PR and it will be summarized by dose level and overall.
Number of Patients with Treatment-related Adverse Events (AEs) and Serious AEs (SAEs) | Recorded at all study visits: weekly (every 7 +/- 2 days) while on treatment and at safety follow-up (35 +/- 5 days post-last dose) or early termination visit (at time of withdrawal).
  (CTCAE) Scale, Version 4.0 for AE grading.
  * Grade 3 neutropenia lasting for ≥ 7 days or granulocyte colony-stimulating factor (G-CSF) administered.
  * Grade 3 thrombocytopenia.
  * Grade 3 treatment-related hyperlipidemia or hypothyroidism
  * Grade 3 study treatment-related non-hematologic toxicity
Pharmacokinetic Parameters | Sampling through 24 hours post end-injection of pralatrexate in cycle 1 dose 1 (week 1) and cycle 1 dose 3 (week 3).
  This was collected during the dose-finding stage of the study. PK sampling is not included in the cohort expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Sharma, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (5):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Ospedale Sant'Orsola - Policlinico Sant'Orsola, Bologna, Italy